CLINICAL TRIAL: NCT01441024
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Study of DAS181 in Patients With Parainfluenza Infection
Brief Title: DAS181 in Patients With Parainfluenza
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 110205; 11-I-0205
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2014-02-27

CONDITIONS: Parainfluenza Infection
Keywords: Immunocompromised; Respiratory Tract Disease; Viral Shedding; Fever; Pharmacokinetics; Parainfluenza Infection; Flu
MeSH Terms: conditions — Paramyxoviridae Infections; Respiratory Tract Diseases; Fever; Influenza, Human | interventions — oplunofusp

ARMS (2):
- 1 (Experimental): DAS181
  Interventions: Drug: DAS181
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DAS181 — 20 mg per day of DAS181-FO3 for 5 days
  Arms: 1
Other: Placebo — 20 mg per day of Lactose for 5 days
  Arms: 2

SUMMARY:
Background:

- Parainfluenza is a virus that can cause infections in people. Most people infected with this virus have mild symptoms including fever, cough, red eyes, or runny nose (a common cold). Some people, especially those with a weakened immune system, get very sick from this virus. They may have difficulty breathing or develop lung infections. Currently, there are no specific treatments for parainfluenza. However, a drug called DAS181 may make the virus go away faster. Researchers are interested in testing DAS181 to see if it is safe and effective against parainfluenza.

Objectives:

- To test the safety and effectiveness of DAS181 as a treatment for parainfluenza.

Eligibility:

- Individuals at least 18 years of age who have the parainfluenza virus and have developed symptoms within the past 10 days.

Design:

* Participants will be screened with a physical exam, medical history, and questions about symptoms and activity levels. Participants will also have a lung function test and provide blood and nasal fluid samples.
* DAS181 is an inhaled medication, and everyone will receive a study medication inhaler. Participants will receive either DAS181 or a placebo through the inhaler. They will take it once every day for 5 days.
* Participants will have monitoring visits on days 2, 4, 7, 10, 14, and 28 to provide blood and nasal fluid samples and have a lung function test.
* Participants who still have the virus in their system on Day 28 will return to the clinic on Day 42 for more tests. Participants who still have the virus in their system on Day 42 will return to the clinic on Day 56 for more tests.
* Participants will have followup visits 6 months and 1 year after the start of the study.

DETAILED DESCRIPTION:
Parainfluenza virus (PIV) infections cause considerable morbidity in the immunocompromised population. In the immunocompetent population, PIV is usually self-limited, but can cause more severe disease including pneumonia and tracheobronchitis in adults, and croup and bronchiolitis in young children. DAS181, an inhaled sialidase, cleaves the binding site of PIV from respiratory mucosal cells limiting the ability of PIV to infect new cells. This may improve outcomes in patients with PIV infections.

This exploratory randomized double-blind Phase 2 study will assess the safety and tolerability, and explore the efficacy of DAS181 versus placebo for the treatment of parainfluenza. Thirty eligible patients diagnosed with parainfluenza will be randomized in a 2:1 allocation to receive either DAS181-F02 formulation (10 mg times 5 days) or placebo. Subjects will be followed on Study Days 0, 2, 4, 7, 10, 14, 28, 180, and 365 with a series of clinical, pulmonary function, functional status, virologic, and safety assessments.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age greater than or equal to 18 years
  2. Positive culture, DFA, PCR or other clinical assay for parainfluenza
  3. Symptomatic upper or lower respiratory tract disease (e.g., pharyngitis, cough, tracheobronchitis, bronchiolitis, pneumonia). Fever alone is not sufficient.
  4. Onset of illness within the last 10 days
  5. Females who are able to become pregnant (i.e., are not postmenopausal, have not undergone surgical sterilization, and are sexually active with men) must agree to use at least 2 effective forms of contraception from the date of informed consent through Study Day 28 of the study. At least 1 of the methods of contraception should be a barrier method
  6. Willingness to have samples stored

EXCLUSION CRITERIA:

1. Known hypersensitivity to DAS181 or any of its components
2. Women who are pregnant (positive serum or urine pregnancy test), who are attempting to become pregnant, or who are breast-feeding
3. Mechanical ventilation, acute respiratory distress, or otherwise unable to tolerate the drug delivery device (Cyclohaler)
4. Allergy or history of allergy to milk or lactose
5. Previous or current history of asthma or chronic obstructive pulmonary disease (COPD) requiring daily medication
6. Any significant findings in the patient s medical history or physical examination that, in the opinion of the investigator, would affect patient safety or compliance with the dosing schedule

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07-14; Primary Completion 2014-02-27 (Actual); Study Completion 2014-06-30 (Actual)

PRIMARY OUTCOMES:
Number patients with at least 1 grade 3/4/SAE that are possibly, probably, or definitely related to the study product by Study Day 28. | study day 28

SECONDARY OUTCOMES:
Virologic Endpoints: Viral shedding by qualitative PCR or culture. | 1 year
Clinical Endpoints: Clinical symptoms, Fever, Radiographic evidence of lower tract disease by CT (if obtained clinically), Death, Hospitalization, Use of supplemental oxygen. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Davey, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)

REFERENCES:
- [Background] Henrickson KJ. Parainfluenza viruses. Clin Microbiol Rev. 2003 Apr;16(2):242-64. doi: 10.1128/CMR.16.2.242-264.2003. PMID 12692097
- [Background] Weintrub PS, Sullender WM, Lombard C, Link MP, Arvin A. Giant cell pneumonia caused by parainfluenza type 3 in a patient with acute myelomonocytic leukemia. Arch Pathol Lab Med. 1987 Jun;111(6):569-70. PMID 3034189
- [Background] Apalsch AM, Green M, Ledesma-Medina J, Nour B, Wald ER. Parainfluenza and influenza virus infections in pediatric organ transplant recipients. Clin Infect Dis. 1995 Feb;20(2):394-9. doi: 10.1093/clinids/20.2.394. PMID 7742447